CLINICAL TRIAL: NCT01962454
Title: A Pilot Study in Healthy Male Volunteers to Evaluate a Skeletal-Muscle Microbiopsy Technique for Suitability of Use With Dynamic Proteomic Measurement
Brief Title: A Study to Evaluate a Skeletal-muscle Microbiopsy Technique With Dynamic Proteomic Measurement in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 200030
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cachexia
Keywords: muscle mass; dynamic proteomics; Duke University; Microbiopsy; D2O; testosterone; skeletal muscle
MeSH Terms: conditions — Cachexia | interventions — testosterone enanthate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Run-in Phase: All participants will receive oral deuterated water (D2O) for 3 weeks prior to the Treatment Phase of the study. The participants will consume 50mL 70% D2O three times per day (TID) for 7 days, followed by a 50ml 70% D2O dose twice daily (BID) for the next 2 weeks. Treatment Phase: Subjects will receive testosterone matching placebo IM injection one per week and 50 mL 70% D2O dose BID for 3 weeks.
  Interventions: Drug: Deuterated Water; Drug: Testosterone enanthate
- Arm 2 (Placebo Comparator): Run-in Phase: All participants will receive oral D2O for 3 weeks prior to the Treatment Phase of the study. The participants will consume 50 mL 70% D2O TID for 7 days, followed by a 50mL 70% D2O dose BID for the next 2 weeks. Treatment Phase: Subjects will receive testosterone IM injection one per week and 50 mL 70% D2O dose BID for 3 weeks
  Interventions: Drug: Deuterated Water; Drug: Placebo to match testosterone enanthate

INTERVENTIONS:
Drug: Deuterated Water — D2O 70% will be supplied as clear liquid, provided in 50 millilitre (mL) unit dose vials; administered per orally.
Drug: Testosterone enanthate — Testosterone enanthate 125mg injection will be supplied as colorless to pale yellow liquid; administered intramuscular (IM).
  Arms: Arm 1
Drug: Placebo to match testosterone enanthate — Placebo to match testosterone enanthate 0.625 mL injection will be supplied as greenish yellow, bright and clear oily liquid; administered intramuscular (IM).
  Arms: Arm 2

SUMMARY:
This is a single-blind, randomized placebo-controlled, parallel study, where the study volunteers will be blinded to testosterone/placebo treatment. This study will test a relatively new, less invasive method for collecting muscle tissue to determine if this method is appropriate for collecting muscle samples for the assessment of the fractional synthetic rates (FSR) of muscle-derived proteins. This study will also investigate whether the FSR of proteins may serve as early biomarkers for muscle anabolism, a known anabolic agent (testosterone) will be administered to healthy, elderly male subjects over a 3 week period. The fractional synthetic rate of several muscle-derived proteins will be analyzed at Baseline and during the period of testosterone treatment using deuterium labelling of these proteins by the incorporation of deuterium from deuterated water (D2O).

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 60-75 of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Ambulatory outside of home, stable chronic conditions allowed (if no clinically significant changes or major medication adjustments in previous 3 months) such as hypertension and/or dyslipidemia. Subjects must be able to satisfactorily complete each lower extremity 1-repetition maximum leg press assessment.
* Body weight >=50 kilogram and body mass index within the range 20 - 34 kilogram per square meter (inclusive)
* Renal clearance >= 45 milliliter per minute based on estimated Glomerular Filtration Rate (eGFR) calculated by the abbreviated MDRD equation, using serum creatinine and demographic data obtained at Screening.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* ALT, alkaline phosphatase and bilirubin =< 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Averaged corrected QT interval (QTc) values of 3 electrocardiograms separated by a 3-5 minute period: Bazett's QTc (QTcB) or Fridericia's QTc (QTcF) < 460 msec; or QTcB or QTcF < 480 msec in subjects with Partial Bundle Branch Block.

Exclusion Criteria:

* Subjects with a history of clinically significant endocrine, gastrointestinal, cardiovascular, neurological, haematological, immunological, renal, respiratory, vertigo, dizziness, prostate enlargement, or genitourinary abnormalities or diseases
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of muscular or neuromuscular disease such as multiple sclerosis, myasthenia gravis, muscular dystrophy, amyotrophic lateral sclerosis, stroke or transient ischemic attack
* Hospitalization in the past 6 months
* Current or recent use of ACE-inhibitors and/or systemic steroids
* Diabetes (Type 1, Type 2)
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the local anaesthetics, study diagnostic reagents, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of bleeding disorder, including thrombocytopenia and other coagulopathies, or current use of anti-coagulants.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus antibody.
* Electrolytes - Sodium more than +-5 milliequivalent per liter (mEq/L) outside the normal reference range, Potassium or Calcium more than 10% outside the normal reference range (<0.9 x lower limit of normal [LLN] or >1.1 x ULN)
* Metabolic - Glucose more than 10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN) or Total Cholesterol > 240 milligram per deciliter
* Muscle - creatine phosphokinase >2.0 x ULN
* Hematology - Hemoglobin, White blood cells, Neutrophils, or Platelets more than 10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN)
* A pro time/prothrombin time test (PT/PTT) outside the normal reference range for the assay.
* Prostate Specific Antigen (PSA) >=3.0 nanogram per milliliter
* Significant prostate enlargement upon clinical examination.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first deuterated water (D2O) dosing day from the Run-in Phase in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first D2O dosing day in the Run-in Phase.

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in muscle derived protein synthesis rate | Baseline and Day 21
  Muscle protein synthesis will be assessed by measuring the fractional synthetic rate of muscle-derived proteins in both muscle biopsy samples and in blood after subjects have ingested deuterated water. The FSR of several muscle-derived proteins will be analyzed at baseline and during the period of testosterone treatment using deuterium labelling of these proteins by the incorporation of deuterium from D2O.

SECONDARY OUTCOMES:
Change from Baseline in lower extremity strength using the 1-repetition maximum (1-RM) leg strength, FSRs from muscle proteins derived from muscle biopsies and serum samples | Baseline, Day 7, 14, and 21
  Lower extremity strength will be measured as the 1-RM on a leg press device. Strength will be measured at baseline (Day 1, prior to start of testosterone) and at study end (Day 21). The FSR of several muscle-derived proteins will be analyzed at Baseline and during the period in both muscle biopsy samples and in blood after subjects have ingested deuterated water.
Changes in FSR in muscle and serum derived muscle proteins | Baseline, Day 7, 14, and 21
  The FSR of several muscle-derived proteins will be analyzed at Baseline and during the period in both muscle biopsy samples and in blood after subjects have ingested deuterated water.
Number of biopsy samples required to obtain desired collection weight | Baseline, Day 7, 14, and 21
Number of participants with biopsy-related adverse events | Upto Week 7

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Durham, North Carolina, United States

REFERENCES:
- See also: Results for study 200030 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200030?search=study&b'search_terms=200030'#rs